CLINICAL TRIAL: NCT05102071
Title: Clinical and Economic Impact of 2nd Line Initiation of Empagliflozin After Metformin, as Compared to 2nd Line Initiation of Sulfonylurea After Metformin in Patients With Type 2 Diabetes and Cardiovascular Disease
Brief Title: Clinical Outcomes and Healthcare Cost and Resource Utilization (HCRU) in Patients With Type 2 Diabetes and Cardiovascular Disease on 2nd Line Empagliflozin Versus 2nd Line Sulfonylureas
Status: Withdrawn | Type: Observational
Why Stopped: Study was canceled because database sample size was inadequate.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0262
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — empagliflozin; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment with empagliflozin: as add-on therapy with metformin
  Interventions: Drug: empagliflozin; Drug: metformin
- Treatment with a sulfonylurea: as add-on therapy with metformin
  Interventions: Drug: metformin; Drug: sulfonylurea

INTERVENTIONS:
Drug: empagliflozin — empagliflozin
  Groups: Treatment with empagliflozin
Drug: metformin — metformin
Drug: sulfonylurea — sulfonylurea
  Groups: Treatment with a sulfonylurea

SUMMARY:
Evaluation of clinical outcomes (specifically cardiovascular outcomes like hospitalization for heart failure), and healthcare cost, and resource utilization, among patients on empagliflozin as an add-on therapy to metformin versus patients on sulfonylureas as an add-on therapy to metformin in patients with Type 2 Diabetes (T2D) and Cardiovascular Disease (CVD).

ELIGIBILITY:
Inclusion criteria:

* Prevalent metformin use + initiation of empagliflozin OR prevalent metformin use + initiation of sulfonylurea
* ≥18 years of age at index date during study observation
* ≥1 inpatient and/or ≥ 2 outpatient claims denoting T2D diagnosis (in any position) in the 12 months prior to index date
* ≥1 inpatient and/or ≥2 outpatient claims denoting CVD (in any position) diagnosis in the 12 months prior to index date
* ≥2 months post-index date
* ≥12 months of no exposure to T2D medications in the pre-index period (excluding metformin in both arms)
* ≥12 months of continuous enrolment prior to index date

Exclusion criteria:

* Diagnosis of Type 1 Diabetes, secondary, or gestational diabetes in the 12 months prior to index date
* Diagnosis of severe comorbidities including malignancy, end-stage renal disease, human immunodeficiency virus, Hepatitis C infection, or organ transplant in the 12 months prior to index date
* Admission to nursing home in the 12 months prior to index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 Diabetes (T2D) and Cardiovascular Disease (CVD).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of first hospitalization for congestive heart failure (HHF) | up to 5 years and 3 months

SECONDARY OUTCOMES:
Hospitalizations | up to 5 years and 3 months
Emergency department (ED) visits | up to 5 years and 3 months
Length of stay | up to 5 years and 3 months
Number of filled drugs | up to 5 years and 3 months
Outpatient visits | up to 5 years and 3 months
All cause cost | up to 5 years and 3 months
  total cost of care, divided by medical (inpatient costs, outpatient costs, emergency costs) and pharmacy costs (all reported in Per Patient Per Month (PPPM) costs)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim Pharmaceuticals Inc, Ridgefield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com